CLINICAL TRIAL: NCT00774436
Title: A Phase II Study of Focal Cryoablation in Low-Risk Prostate Cancer
Brief Title: Study of Focal Cryoablation in Low-Risk Prostate Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 08-118
Record Dates: First submitted 2008-10-15; First posted 2008-10-17 (Estimated); Last update posted 2019-07-29 (Actual); Status verified 2018-10

CONDITIONS: Prostate Cancer
Keywords: focal cryotherapy; low-risk prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms

ARMS (1):
- Patients scheduled to receive Focal Cryotherapy (Experimental): After enrollment, patients will undergo a repeat transrectal ultrasound- guided prostate biopsy (minimum of 12 cores) to confirm the low-risk nature of their cancer. For study purposes, patients must meet the original entry crieteria on this repeat biopsy. If the patient meets the repeat-biopsy enrollment criteria, they will be treated with focal cryotherapy, meaning cryoablation of the regions of the prostate containing cancer. Efficacy is defined as all negative biopsy cores at the site of the focal ablation on a repeat transrectal biopsy 6 months after cryoablation. At baseline (prior to the re-staging biopsy), 3 months after focal cryotherapy, and at 6 months after focal cryotherapy (prior to the repeat prostate biopsy used to define efficacy), the patient will complete quality of life questionnaires as standard for all patients in the Urology Service.
  Interventions: Procedure: focal cryotherapy

INTERVENTIONS:
Procedure: focal cryotherapy — Those men meeting the re-staging biopsy criteria will subsequently be treated with focal cryotherapy. Clinical follow-up visits will be scheduled at 6 + 2 weeks, 3 + 1 months and 6 + 1 months after focal cryotherapy, at which time, a digital rectal examination and PSA test will be performed. Standard quality-of-life questionnaires, are completed by all patients treated by the Urology Service (whether on not they are treated on an IRB protocol).

SUMMARY:
The purpose of this study is to find out if men, with low-risk prostate, can have the small amount of cancer within their prostate removed by freezing, called Focal Cryoablation or Cryotherapy.

ELIGIBILITY:
A two-step consenting process will be in place for all patients being enrolled to this study. The two-step method is necessary because all patients being enrolled will need to have a repeat transrectal biopsy after meeting the initial study requirements. The two step consent process would enroll patients considering focal cryotherapy into the initial part of the study (QOL assessment at baseline, PCA3 test, and repeat biopsy); those deemed eligible after the re-staging biopsy would be consented to participate in the remainder of the study (focal cryotherapy, QOL studies, repeat biopsy at 6 months for efficacy, PCA3 test).

First Step Enrollment

Inclusion Criteria:

* Men ≥ 21 years of age with a life expectancy estimated to be > 10-years.
* Diagnosis of adenocarcinoma of the prostate and confirmed by MSKCC review
* No prior treatment for prostate cancer
* ECOG performance status of 0 or 1
* Prostate cancer clinical stage T1c-T2a
* PSA < 10ng/mL (this will be the PSA level prompting the prostate biopsy)
* Prostate Size <60 cc on transrectal ultrasound
* Exclusion Criteria:
* Medically unfit for anesthesia
* Histology other than adenocarcinoma
* Men who have received any hormonal manipulation (antiandrogens; LHRH agonists) within the previous 6 months
* Men who are currently receiving anticoagulant drugs (e.g.: Coumadin, warfarin)

Second Step Enrollment

Inclusion Criteria:

* Repeat transrectal prostate biopsy that must meet the following parameters:
* Minimum of 12 biopsy cores
* No Biopsy Gleason grade 4 or 5
* Unilateral cancer (only right-sided or left-sided, not bilateral)
* No more than 50% cancer in any one biopsy core
* No more than 25% of cores containing cancer

Exclusion Criteria:

* Medically unfit for anesthesia
* Histology other than adenocarcinoma
* Men who have received any hormonal manipulation (antiandrogens; LHRH agonists) within the previous 6 months
* Men who are currently receiving anticoagulant drugs (e.g.: coumadin, warfarin)

Min Age: 21 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2008-10-14 (Actual); Primary Completion 2019-07-23 (Actual); Study Completion 2019-07-23 (Actual)

PRIMARY OUTCOMES:
To assess the local oncologic efficacy of focal cryoablation in men with low-risk, clinically localized prostate cancer, as measured by the ability to obtain all negative biopsy cores at the site of focal ablation of the cancer. | conclusion of the study

SECONDARY OUTCOMES:
To evaluate the change from baseline in quality-of-life indicators following focal cryoablation in patients with low-risk localized prostate cancer. | conclusion of the study
To evaluate treatment related tissue changes with ultrasound imaging | prior to performing the biopsy
  Ultrasound examination of the prostate performed at the time of biopsy procedures will be include archiving of 3D digital images to allow post-hoc analysis of the images to assess for tissue changes that may be characterized with imaging software.
To evaluate treatment related tissue changes with ultrasound imaging | at the 6-8 month patient office visit
  Ultrasound examination of the prostate performed at the time of biopsy procedures will be include archiving of 3D digital images to allow post-hoc analysis of the images to assess for tissue changes that may be characterized with imaging software.

CONTACTS AND LOCATIONS:
Overall Officials: James Eastham, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan-Kettering Cancer Center, New York, New York, United States

REFERENCES:
- See also: Memorial Sloan-Kettering Cancer Center — http://www.mskcc.org